CLINICAL TRIAL: NCT02193100
Title: PRE AND POST TREATMENT METABOLOMIC ANALYSIS OF LEUKEMIA: A Translational Clinical Trial of the Brown Cancer Center
Status: Withdrawn | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: BCC-BMT-13 Leuk Metabolomics
Record Dates: First submitted 2014-06-12; First posted 2014-07-17 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2016-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 13C-glucose: experimental (13C-glucose)
- No glucose: control (no glucose)

SUMMARY:
To characterize the metabolism of glucose by the leukemic cells in patients with leukemia before and after initial chemotherapy.

To compare the metabolism of glucose by leukocytes in healthy volunteers and leukemic cells in leukemic patients.

DETAILED DESCRIPTION:
To characterize glycolytic metabolism in patients as demonstrated in leukemic cells and serum metabolite analysis after C13-glucose administration at strategic time points of treatment.

To detect and measure 13C-labeled metabolic markers which may be present in the serum and urine of leukemic patients.

To characterize glycolytic metabolism in patients as demonstrated in leukemic cells and serum metabolite analysis after C13-glucose administration at strategic time points of treatment.

To detect and measure 13C-labeled metabolic markers which may be present in the serum and urine of leukemic patients.

ELIGIBILITY:
Inclusion Criteria for Leukemia Subjects:

* Each of the criteria in the following section must be met in order for a patient to be eligible for enrollment.
* Only patients with clinically diagnosed or histologically diagnosed leukemia will be eligible to participate in this non-therapeutic study.
* All patients must have measurable quantities of leukemic blasts on peripheral blood detected with a CBC.
* No history of diabetes for the experimental group or the control group.
* Patients with known hepatitis C or HIV (AIDS) are excluded.
* Patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.

Inclusion Criteria forHealthy Subjects:

* Subjects must have no known prior history of cancer or malignant blood disorders. -Where possible, follow up will be carried out to verify that no cancer has developed since the blood collection. This will be done by a phone call performed one month from sample to ask if new medical conditions have arisen.
* Subjects must have WBC, RBC, and platelet counts within normal range on CBC.
* Subjects with known hepatitis C or HIV (AIDS) are excluded.
* No history of Diabetes
* At least 30 years of age
* Preferably be fasting for 12 hours (minimum 8 hours) prior to enrollment
* Patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* None listed in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Leukemia Subjects-clinically diagnosed or histologically diagnosed leukemia Healthy Subjects-no record of diagnosed cancer or hematologic disorders
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Metabolic characteristics of leukemic cells from blood and urine samples using nuclear magnetic resonance spectroscopy (NMR) | Baseline up to 6 months post treatment
  Blood and urine samples will be taken before and after chemotherapy treatment for up to 6 months post treatment and analyzed for metabolic substances using nuclear magnetic resonance (NMR) spectroscopy with intergraded hyphenated mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- James Graham Brown Cancer Center-University of Louisville, Louisville, Kentucky, United States